CLINICAL TRIAL: NCT07312162
Title: Multilevel Determinants of Socioeconomic Disparities in Geographic Late-Stage Hepatocellular Carcinoma Hotspots
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19PS-21-7; NCI-2024-03737 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19PS-21-7 (Other: USC / Norris Comprehensive Cancer Center); K23MD016963 (NIH); P30CA014089 (NIH)
Record Dates: First submitted 2024-05-20; First posted 2025-12-31 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Participants complete surveys, have their medical records reviewed, and may complete an interview on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates barriers to early detection of liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify individual-level social and clinical determinants of socioeconomic disparities in late stage Hepatocellular Carcinoma (HCC) burden with a prospective survey of patients with incident HCC. II. To qualitatively explore the multilevel barriers to completion of the early detection pathway for HCC in low socioeconomic status (SES) populations.

OUTLINE: This is an observational study.

Participants complete surveys, have their medical records reviewed, and may complete an interview on study.

ELIGIBILITY:
Inclusion Criteria:

* * Adults (18+)

  * New diagnosis of HCC
  * Able to provide informed consent

Additional criteria:

* Must complete survey
* Residential address in a late stage hotspot
* Medicaid insurance or uninsured
* English, Spanish and Chinese speakers

Exclusion Criteria:

* * Residence outside of Los Angeles County

  * Non-HCC liver tumors
  * Incarcerated patients
  * Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (18+ years of age) of all stages with a diagnosis of HCC defined by guideline-based radiographic findings on cross-sectional imaging and/or histopathology
Sampling Method: Non-Probability Sample
Enrollment: 730 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Social determinants of health | Up to 4 years
  Patient social determinants of health-related needs will be measured through a health questionnaire created for the study. The patient can respond yes or no to having a lack of transportation to and from appointments. The patient is given a scale of never true, sometimes true and often true for questions regarding food insecurity. The patient can indicate that they do or do not have housing today (or choose not to answer), and they can indicate how many times they moved in the last year as 0, 1, or 2+. For the remaining questions regarding housing, paying for utilities, paying for medications, unemployment, education and child or family care, the patient can respond yes, no or choose not to answer. Responses of yes indicate the patient has a need, and no indicates that they do not have a need.
Barriers to completion of the early detection pathway for liver cancer | Up to 4 years
  For assessment we will conduct semi-structured interviews with key stakeholders, including low-income patients with liver cancer, providers in an interconnected safety net system, and community leaders of hotspot neighborhoods.

CONTACTS AND LOCATIONS:
Overall Officials: Kali Zhou, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States